CLINICAL TRIAL: NCT06623110
Title: A Phase 2 Study of Intralesional RP2 as Immunoprevention for High-Risk Oral Precancerous Disease (INTERCEPT)
Brief Title: Phase II Study of RP2 as Immunoprevention in High-Risk Oral Precancerous Disease
Acronym: INTERCEPT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glenn J. Hanna (Other)
Collaborators: Replimune Inc. (Industry)
Responsible Party: Sponsor-Investigator, Glenn J. Hanna, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-383
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: High-Risk Oral Precancerous Disease
Keywords: High-Risk Oral Precancerous Disease; Oral Precancerous Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP2 Injection (Experimental): Enrolled participants will complete the following:
  * A 3 subject safety run-in will be conducted with participants enrollment staggered. If > 1 subject experiences a grade 4-5 adverse event (AE), study enrollment will pause for review by PI and study sponsor. If there are 0 grade 4-5 AEs, enrollment will proceed.
  * Baseline in-clinic visit with assessments, oral mucosal punch biopsy, and RP2 injection (week 1).
  * In-clinic visits on weeks 3, 5, 7, 8, 9, 11, 13, 15, and 16.
  * RP2 injections on weeks 1, 3, 5, 7, 9, 11, 13, and 15.
  * Repeat oral mucosal punch biopsy at week 8.
  * Follow up: every 3 months for up to 2 years.
  Interventions: Biological: RP2 Injection

INTERVENTIONS:
Biological: RP2 Injection — Genetically modified live HSV-1 virus, 3.0 mL single-use glass vials, via intralesional (into a lesion) injection per protocol.

SUMMARY:
The goal of this study is to understand the safety, tolerability, and potential efficacy of an injected immune therapy called RP2 to treat oral precancer conditions and prevent progression to an oral cancer.

The name of the study drug involved in this study is:

-RP2 (a genetically modified live Herpes Simplex V-1 strain)

DETAILED DESCRIPTION:
This is a single-arm, open-label, single-center phase 2 study evaluating RP2 as a therapy for participants with high-risk oral precancerous diseases (OPDs).

RP2 is a herpes simplex virus (a viral infection commonly known as the "cold sore virus") that has been changed to grow in and destroy cancer cells and to activate (turn on) the human immune system to attack the cancer cells. RP2 is made using herpes simplex virus type-1 (HSV-1) viral carrier which has been changed such that it is unlikely to cause human disease

The U.S. Food and Drug Administration (FDA) has not approved RP2 as a treatment for high-risk oral precancerous disease.

The study procedures for this research study include a screening visit to determine eligibility, in-clinic visits, blood tests, urine tests, and mucosal punch biopsy,

Participants will receive the study drug every 2 weeks and will be followed for up to 2 years.

It is expected that up to 25 people will take part in this research study.

Replimune, Inc. is supporting this study by supplying the drug, RP2, and providing funding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of high-risk OPD defined by any of the following:

  * Proliferative leukoplakia (PL)
  * Localized leukoplakia showing at least moderate dysplasia not treated with surgery
  * Erythroplakia (regardless of dysplasia)
  * High-risk LOH profile: 9p21 or CDKN2A or MTAP loss; regardless of personal oral cancer history
  * Any degree of dysplasia with a known TP53 mutation
  * A history of treated stage 1 or 2 (AJCC 2017 8th edition) HNSCC with at least moderate dysplasia at the resection margins or known 9p21 loss or a known TP53 mutation
* No evidence of head and neck cancer recurrence within the last 3 months (if applicable).
* Willing to provide blood and tissue for diagnostic biopsies.
* At least one target injectable measurable lesion ≥1 cm in longest diameter that can be followed.
* Any smoking history is permitted. While discouraged, patients are permitted to continue tobacco use while on the study.
* Age 18 years or older at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Participant must have normal marrow function and coagulation profile as defined within 21 days prior to study registration:

  * absolute neutrophil count ≥1,000/mcL
  * hemoglobin ≥9 g/dL
  * platelets ≥75,000/mcL, and (d) PT/INR <2.5, and (e) aPTT <1.5x ULN.
* Women of childbearing potential (WOCBP) must agree to use appropriate method(s) of contraception. WOCBP and men should plan to use an adequate method to avoid pregnancy for 90 days after the last dose of RP2. WOCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Serum or urine BhCG testing is required within 24 hours of initial RP2 dosing.

Exclusion Criteria:

* Prior treatment with an oncolytic virus therapy.
* Systemic infection requiring intravenous (IV) antibiotics.
* Requires chronic use of systemic (oral or IV) antivirals with known antiherpetic activity (e.g. acyclovir or valacyclovir).
* Active significant herpetic infections or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis). Patients with sporadic cold sores may be enrolled provided they are asymptomatic at the time of starting RP2.
* Known acute or chronic hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or acute or chronic hepatitis C virus (defined as HCV RNA [qualitative] is detected). Note: Patients who have been effectively treated are eligible for enrollment. Patients must be negative for HBsAg and HCV RNA.
* Known human immunodeficiency virus (HIV) infection. Note: Testing for HIV is not required unless mandated by local health authority or clinically indicated.
* A history of a prior stage III (T1-2N1, T3N0) or IV (T1-3N2, T4N0) invasive head & neck squamous cell carcinoma treated with surgery and/or radiation with or without chemotherapy.
* Patients cannot be on long-term (>4 weeks) corticosteroids at doses exceeding prednisone 20 mg daily (or its equivalent) at the time of enrollment.
* A personal history of hematopoietic stem cell (bone marrow) or solid organ transplant.
* A personal history of other active malignancies, with exceptions including (but not limited to): non-melanomatous skin cancers, low-risk prostate adenocarcinoma on active surveillance, or treated cancers in remission for the last 2 years.
* Significant bleeding event within the last 6 months that places the patient at risk for bleeding due to the injection procedure based on Investigator assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response | Up to 1 year
  The best overall response is the best response recorded from the start of the treatment until disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Responses do not require confirmation. Complete response (CR) is complete disappearance of all target lesions. Partial response (PR) is at least 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Adverse Event Rate | Up to 1 year
  Adverse event rate is defined as the proportion of participants experiencing adverse. Adverse events will be classified and graded according to CTCAE5.0.
Median Cancer-free Survival (CFS) | Up to 1 year
  Cancer-Free Survival (CFS) is defined as the time from study registration to development of a biopsy-proven invasive oral cancer (oral squamous cell carcinoma or OSCC) or time to a primary, recurrent, or secondary biopsy-proven invasive head and neck cancer diagnosis (squamous cell carcinoma of the head and neck) or death due to any cause. Participants alive without disease progression or recurrence (of invasive oral cancer) are censored at date of last disease evaluation.
Median Overall Survival (OS) | Up to 3 years
  Overall Survival (OS) based on Kaplan-Meier method is defined as the time from registration to death due to any cause, or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu